CLINICAL TRIAL: NCT03601585
Title: Evaluation of the Effectiveness of Fibrous Foods, Sugar-free Gomes and Rolly Brush® in the Dental Biofilm Removal: A Randomized, Double Masked Clinical Trial
Brief Title: Evaluation of the Effectiveness of Fibrous Foods, Sugar-free Gomes and Rolly Brush® in the Dental Biofilm Removal
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Olga Flecha, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: self-cleaning
Record Dates: First submitted 2018-07-10; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Self Cleaning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rolly Brush (Experimental): Chew for 1 minute
  Interventions: Device: Comparison of dental biofilm removal.
- Chewing gum (Experimental): Chew for 1 minute
  Interventions: Device: Comparison of dental biofilm removal.
- Apple (Experimental): Chew for 1 minute
  Interventions: Device: Comparison of dental biofilm removal.
- Brush (Active Comparator): brush for 1 minute
  Interventions: Device: Comparison of dental biofilm removal.

INTERVENTIONS:
Device: Comparison of dental biofilm removal. — Comparison of the use of 4 methods for dental biofilm removal

SUMMARY:
The objective of this study was to evaluate the efficacy of three methods for removal of dental biofilm when compared to dental toothbrushing control. Twenty patients were diagnosed and randomized into four groups according to the method tested: 1) apple 2) Rolly Brush 3) chewing gum and 4) brushing control. Subjects were evaluated four times according to the method used. All were evaluated before performing any method and after using each of the four methods separately. The patient's evaluation interval was 24 hours between the use of the methods. In the first stage, they underwent a clinical examination in which the needs of supragingival scraping or definitive restorations and prophylaxis were detected. After this step, all methods of oral hygiene and the consumption of fibrous foods and chewing gum were suspended for twenty-four hours. In the second stage, with a minimum of twenty-four hours after the first, volunteers received approximately 10 ml of basic fucsin to perform a mouthwash. The dental examination was then carried out for measurement on each dental surface and the plaque index was recorded on each surface. In the latter, four evaluations were performed with at least a 24-hour interval until the patients used the four methods

ELIGIBILITY:
Inclusion Criteria:

* Good periodontal health
* Minimum of eight occlusal surfaces of premolars and molars hygienic

Exclusion Criteria:

* Less than eight occlusal surfaces
* Use of orthodontic appliance
* Use of dental prosthesis

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Plaque index | 3 months
  Comparison of the Quigley-Hein plaque index between the following groups: rolly brush, chewing gum, a, apple, brush.

CONTACTS AND LOCATIONS:
Locations (1):
- Periodontics Clinic, Department of Dentistry, Diamantina, Minas Gerais, Brazil